CLINICAL TRIAL: NCT06294808
Title: Predicting Survival After Surgical Resection for the Entire Spectrum of Anatomically Resectable HCC: a Metroticket Approach
Brief Title: Predicting Survival After Surgical Resection for the Entire Spectrum of Anatomically Resectable HCC
Status: Completed | Type: Observational
Sponsor: National Cancer Centre, Singapore (Other)
Collaborators: Singapore General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-2601
Record Dates: First submitted 2024-02-26; First posted 2024-03-06 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Hepatocellular Carcinoma Resectable
Keywords: Metroticket Approach; Surgical Resection; Hepatocellular Carcinoma (HCC)
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Clinical outcomes after surgical resection in HCC is a continuum and is clearly related to tumor burden but needs better definition. The researchers describe the use of the "metro ticket" approach to analyze surgical outcomes over the whole spectrum of anatomically resectable HCC to define overall survival including intermediate stage tumors (BCLC B). The analysis the researchers provide in this study enables the clinician to select the optimal surgical resection candidate based on robust long term survival data.

In addition, study compares outcome for open surgery vs laparoscopic surgery, survival outcome for viral and non-viral HCC using Albumin-Bilirubin (ALBI) for more comprehensive study result.

On top of that, non-HBV, non-HCV (NBNC) hepatocellular carcinoma (HCC) is generally associated with poorer tumor characteristics. However, it remains unclear whether this leads to worse post-resection survival compared to viral-related HCC. This study evaluates the prognostic impact of viral status and liver function on post-resection survival outcomes between NBNC and viral HCC patients.

This retrospective study also aims to determine if HCC of viral and non-viral etiologies have different clinical outcomes after surgical resection when tumor burden and liver function are considered.

DETAILED DESCRIPTION:
Patients who underwent surgical resection (both open surgery and laparoscopic surgery) for HCC from 1st January 2000 to 30th June 2018 by the joint hepato-pancreato-biliary surgery service at the Singapore Healthcare Group of Hospitals (Singapore General Hospital and the National Cancer Centre Singapore) were retrospectively identified from a prospectively kept institutional database.

The assessment of the size, number of nodules and vascular invasion of HCC were based on pre-operative CT/MRI imaging and pathological assessment of the resected specimens. All resections were histologically confirmed as HCC. Patients with macrovascular invasion and extrahepatic invasion were excluded from analysis as were patients resected for other palliative intents (e.g. ruptured HCC).

ELIGIBILITY:
Inclusion Criteria:

1. Unequivocal diagnosis of Hepatocellular Carcinoma (HCC) by histology
2. Patients who underwent surgical resection for HCC

Exclusion Criteria:

1. Patients who underwent liver resection for other malignancies ie cholangiocarcinoma
2. Patients with HCC who did not undergo liver resection.
3. Patients with HCC who underwent liver transplant.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent surgical resection (both open surgery and laparoscopic surgery) for HCC from 1st January 2000 to 30th June 2018 by the joint hepato-pancreato-biliary surgery service at the Singapore Healthcare Group of Hospitals (Singapore General Hospital and the National Cancer Centre Singapore).
Sampling Method: Non-Probability Sample
Enrollment: 1043 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
5-year mortality. | At least 5 years.
  Time between the respective surgery to the time of death. Bivariate contour plots of 5-year survival probability as a function of X = AFP concentration (ng/mL) and Y = tumor burden index (size of largest nodule + 2*number of nodules) (TBI) were obtained as smoothed contours originating from an empirically-derived bivariate 5-year survival distribution S(X,Y)=1- F(x ≤X,y ≤Y). The function F(x ≤X,y ≤Y) is the empirical, bivariate cumulative distribution of 5-year mortality as a function of X and Y defined over the domain (0<X≤5000,1≤Y≤15) in our patient cohort. All patients in our study cohort were followed up for at least 5 years following respective surgery which allowed estimation of actual all-cause 5-year mortality.
Concordance of pre-operative radiological and post operative surgical specimen. | Through study completion, an average of 3 years.
  The metro ticket modeling was based on tumour size and number of nodules extracted at pre-operative radiological imaging and post surgical pathology assessment. Continuous variables are summarized as mean, standard deviation, 25th and 75th percentiles, median and minimum and maximum. Categorical variables are summarized as counts (N) and percentages (%).
Agreement between TBI calculated from pre-operative imaging versus those obtained from post-surgical pathological assessment. | Through study completion, an average of 3 years.
  Bland-Altman analysis, which is based on a simple but effective graphical approach for evaluating bias and for calculating bounds on the expected magnitude of the individual differences arising between the two measurement methods, is used. A 45° line of identity with scatter plot was produced to display the correlation between the 2 measurements. Bias was evaluated by calculating (d) ̅ the mean difference of the measurements. Limits of agreement, calculated as (d) ̅ ±2sd , where sd is the standard deviation of the individual differences, defined bounds within which 95% of the measurement differences are expected to fall. The B-A plot defines the limits of agreements. B-A analysis is performed using TBI over a wide range, 0 ≤ TBI ≤ 30, and a restricted range focusing on small tumors, 0 < TBI ≤ 6.
Overall survival (OS) stratified on hepatitis status. | Minimum 2 years follow up after Hepatocellular carcinoma resection.
  The time elapsed from the surgical resection to the point of death or the last follow-up, whichever occurred first.
Recurrence-free survival (RFS) stratified on hepatitis status. | Minimum 2 years follow up after Hepatocellular carcinoma resection.
  The time between surgical resection of HCC and its recurrence confirmed via multi-phasic CT or MRI imaging, or last follow-up, whichever occurred first.
Prognostic stratification according to ALBI grade. | Minimum 2 years follow up after Hepatocellular carcinoma resection.
  Overall survival (OS) and Recurrence-free survival (RFS) stratified according to ALBI grade.

CONTACTS AND LOCATIONS:
Overall Officials: Pierce Chow, MD, PhD, Principal Investigator — National Cancer Centre, Singapore
Locations (2):
- Singapore (2):
  - National Cancer Centre, Singapore, Singapore
  - Singapore General Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ferlay J, Shin HR, Bray F, Forman D, Mathers C, Parkin DM. Estimates of worldwide burden of cancer in 2008: GLOBOCAN 2008. Int J Cancer. 2010 Dec 15;127(12):2893-917. doi: 10.1002/ijc.25516. PMID 21351269
- [Background] Omata M, Lesmana LA, Tateishi R, Chen PJ, Lin SM, Yoshida H, Kudo M, Lee JM, Choi BI, Poon RT, Shiina S, Cheng AL, Jia JD, Obi S, Han KH, Jafri W, Chow P, Lim SG, Chawla YK, Budihusodo U, Gani RA, Lesmana CR, Putranto TA, Liaw YF, Sarin SK. Asian Pacific Association for the Study of the Liver consensus recommendations on hepatocellular carcinoma. Hepatol Int. 2010 Mar 18;4(2):439-74. doi: 10.1007/s12072-010-9165-7. PMID 20827404
- [Background] Edge SB, Compton CC. The American Joint Committee on Cancer: the 7th edition of the AJCC cancer staging manual and the future of TNM. Ann Surg Oncol. 2010 Jun;17(6):1471-4. doi: 10.1245/s10434-010-0985-4. PMID 20180029
- [Background] Forner A, Llovet JM, Bruix J. Hepatocellular carcinoma. Lancet. 2012 Mar 31;379(9822):1245-55. doi: 10.1016/S0140-6736(11)61347-0. Epub 2012 Feb 20. PMID 22353262
- [Background] Lim KC, Chow PK, Allen JC, Siddiqui FJ, Chan ES, Tan SB. Systematic review of outcomes of liver resection for early hepatocellular carcinoma within the Milan criteria. Br J Surg. 2012 Dec;99(12):1622-9. doi: 10.1002/bjs.8915. Epub 2012 Sep 28. PMID 23023956
- [Background] Mazzaferro V, Llovet JM, Miceli R, Bhoori S, Schiavo M, Mariani L, Camerini T, Roayaie S, Schwartz ME, Grazi GL, Adam R, Neuhaus P, Salizzoni M, Bruix J, Forner A, De Carlis L, Cillo U, Burroughs AK, Troisi R, Rossi M, Gerunda GE, Lerut J, Belghiti J, Boin I, Gugenheim J, Rochling F, Van Hoek B, Majno P; Metroticket Investigator Study Group. Predicting survival after liver transplantation in patients with hepatocellular carcinoma beyond the Milan criteria: a retrospective, exploratory analysis. Lancet Oncol. 2009 Jan;10(1):35-43. doi: 10.1016/S1470-2045(08)70284-5. Epub 2008 Dec 4. PMID 19058754
- [Background] Bruix J, Sherman M; American Association for the Study of Liver Diseases. Management of hepatocellular carcinoma: an update. Hepatology. 2011 Mar;53(3):1020-2. doi: 10.1002/hep.24199. No abstract available. PMID 21374666
- [Background] Zhong JH, Ke Y, Gong WF, Xiang BD, Ma L, Ye XP, Peng T, Xie GS, Li LQ. Hepatic resection associated with good survival for selected patients with intermediate and advanced-stage hepatocellular carcinoma. Ann Surg. 2014 Aug;260(2):329-40. doi: 10.1097/SLA.0000000000000236. PMID 24096763
- [Background] Lin CT, Hsu KF, Chen TW, Yu JC, Chan DC, Yu CY, Hsieh TY, Fan HL, Kuo SM, Chung KP, Hsieh CB. Comparing hepatic resection and transarterial chemoembolization for Barcelona Clinic Liver Cancer (BCLC) stage B hepatocellular carcinoma: change for treatment of choice? World J Surg. 2010 Sep;34(9):2155-61. doi: 10.1007/s00268-010-0598-x. PMID 20407768
- [Background] Ng KK, Vauthey JN, Pawlik TM, Lauwers GY, Regimbeau JM, Belghiti J, Ikai I, Yamaoka Y, Curley SA, Nagorney DM, Ng IO, Fan ST, Poon RT; International Cooperative Study Group on Hepatocellular Carcinoma. Is hepatic resection for large or multinodular hepatocellular carcinoma justified? Results from a multi-institutional database. Ann Surg Oncol. 2005 May;12(5):364-73. doi: 10.1245/ASO.2005.06.004. Epub 2005 Mar 31. PMID 15915370
- [Background] Yang LY, Fang F, Ou DP, Wu W, Zeng ZJ, Wu F. Solitary large hepatocellular carcinoma: a specific subtype of hepatocellular carcinoma with good outcome after hepatic resection. Ann Surg. 2009 Jan;249(1):118-23. doi: 10.1097/SLA.0b013e3181904988. PMID 19106686
- [Background] Torzilli G, Belghiti J, Kokudo N, Takayama T, Capussotti L, Nuzzo G, Vauthey JN, Choti MA, De Santibanes E, Donadon M, Morenghi E, Makuuchi M. A snapshot of the effective indications and results of surgery for hepatocellular carcinoma in tertiary referral centers: is it adherent to the EASL/AASLD recommendations?: an observational study of the HCC East-West study group. Ann Surg. 2013 May;257(5):929-37. doi: 10.1097/SLA.0b013e31828329b8. PMID 23426336
- [Background] European Association For The Study Of The Liver; European Organisation For Research And Treatment Of Cancer. EASL-EORTC clinical practice guidelines: management of hepatocellular carcinoma. J Hepatol. 2012 Apr;56(4):908-43. doi: 10.1016/j.jhep.2011.12.001. No abstract available. PMID 22424438
- [Background] Ishizawa T, Hasegawa K, Aoki T, Takahashi M, Inoue Y, Sano K, Imamura H, Sugawara Y, Kokudo N, Makuuchi M. Neither multiple tumors nor portal hypertension are surgical contraindications for hepatocellular carcinoma. Gastroenterology. 2008 Jun;134(7):1908-16. doi: 10.1053/j.gastro.2008.02.091. Epub 2008 Mar 8. PMID 18549877
- [Background] Peng ZW, Guo RP, Zhang YJ, Lin XJ, Chen MS, Lau WY. Hepatic resection versus transcatheter arterial chemoembolization for the treatment of hepatocellular carcinoma with portal vein tumor thrombus. Cancer. 2012 Oct 1;118(19):4725-36. doi: 10.1002/cncr.26561. Epub 2012 Feb 22. PMID 22359112
- [Background] Sangro B, Inarrairaegui M, Bilbao JI. Radioembolization for hepatocellular carcinoma. J Hepatol. 2012 Feb;56(2):464-73. doi: 10.1016/j.jhep.2011.07.012. Epub 2011 Aug 2. PMID 21816126
- [Background] Khor AY, Toh Y, Allen JC, Ng DC, Kao YH, Zhu G, Choo SP, Lo RH, Tay KH, Teo JY, Goh BK, Burgmans MC, Irani FG, Goh AS, Chow PK. Survival and pattern of tumor progression with yttrium-90 microsphere radioembolization in predominantly hepatitis B Asian patients with hepatocellular carcinoma. Hepatol Int. 2014 Jul;8(3):395-404. doi: 10.1007/s12072-014-9533-9. Epub 2014 Apr 5. PMID 26202641
- [Background] Mazzaferro V, Regalia E, Doci R, Andreola S, Pulvirenti A, Bozzetti F, Montalto F, Ammatuna M, Morabito A, Gennari L. Liver transplantation for the treatment of small hepatocellular carcinomas in patients with cirrhosis. N Engl J Med. 1996 Mar 14;334(11):693-9. doi: 10.1056/NEJM199603143341104. PMID 8594428
- [Background] Yao FY, Ferrell L, Bass NM, Watson JJ, Bacchetti P, Venook A, Ascher NL, Roberts JP. Liver transplantation for hepatocellular carcinoma: expansion of the tumor size limits does not adversely impact survival. Hepatology. 2001 Jun;33(6):1394-403. doi: 10.1053/jhep.2001.24563. PMID 11391528
- [Background] Chang WT, Kao WY, Chau GY, Su CW, Lei HJ, Wu JC, Hsia CY, Lui WY, King KL, Lee SD. Hepatic resection can provide long-term survival of patients with non-early-stage hepatocellular carcinoma: extending the indication for resection? Surgery. 2012 Nov;152(5):809-20. doi: 10.1016/j.surg.2012.03.024. Epub 2012 Jul 3. PMID 22766361
- [Background] Llovet JM, Bruix J. Systematic review of randomized trials for unresectable hepatocellular carcinoma: Chemoembolization improves survival. Hepatology. 2003 Feb;37(2):429-42. doi: 10.1053/jhep.2003.50047. PMID 12540794
- [Background] Cheng AL, Kang YK, Chen Z, Tsao CJ, Qin S, Kim JS, Luo R, Feng J, Ye S, Yang TS, Xu J, Sun Y, Liang H, Liu J, Wang J, Tak WY, Pan H, Burock K, Zou J, Voliotis D, Guan Z. Efficacy and safety of sorafenib in patients in the Asia-Pacific region with advanced hepatocellular carcinoma: a phase III randomised, double-blind, placebo-controlled trial. Lancet Oncol. 2009 Jan;10(1):25-34. doi: 10.1016/S1470-2045(08)70285-7. Epub 2008 Dec 16. PMID 19095497
- [Background] Oliveri RS, Wetterslev J, Gluud C. Transarterial (chemo)embolisation for unresectable hepatocellular carcinoma. Cochrane Database Syst Rev. 2011 Mar 16;2011(3):CD004787. doi: 10.1002/14651858.CD004787.pub2. PMID 21412886
- [Background] Poon RT, Fan ST, Wong J. Selection criteria for hepatic resection in patients with large hepatocellular carcinoma larger than 10 cm in diameter. J Am Coll Surg. 2002 May;194(5):592-602. doi: 10.1016/s1072-7515(02)01163-8. PMID 12022599
- [Background] Yeh CN, Lee WC, Chen MF. Hepatic resection and prognosis for patients with hepatocellular carcinoma larger than 10 cm: two decades of experience at Chang Gung memorial hospital. Ann Surg Oncol. 2003 Nov;10(9):1070-6. doi: 10.1245/aso.2003.03.072. PMID 14597446
- [Background] Nagano Y, Tanaka K, Togo S, Matsuo K, Kunisaki C, Sugita M, Morioka D, Miura Y, Kubota T, Endo I, Sekido H, Shimada H. Efficacy of hepatic resection for hepatocellular carcinomas larger than 10 cm. World J Surg. 2005 Jan;29(1):66-71. doi: 10.1007/s00268-004-7509-y. PMID 15599739
- [Background] Yamashita Y, Taketomi A, Shirabe K, Aishima S, Tsuijita E, Morita K, Kayashima H, Maehara Y. Outcomes of hepatic resection for huge hepatocellular carcinoma (>/= 10 cm in diameter). J Surg Oncol. 2011 Sep 1;104(3):292-8. doi: 10.1002/jso.21931. Epub 2011 Apr 4. PMID 21465490
- [Background] O'Malley ME, Takayama Y, Sherman M. Outcome of small (10-20 mm) arterial phase-enhancing nodules seen on triphasic liver CT in patients with cirrhosis or chronic liver disease. Am J Gastroenterol. 2005 Jul;100(7):1523-8. doi: 10.1111/j.1572-0241.2005.41814.x. PMID 15984975
- [Background] Shah SA, Tan JC, McGilvray ID, Cattral MS, Cleary SP, Levy GA, Greig PD, Grant DR. Accuracy of staging as a predictor for recurrence after liver transplantation for hepatocellular carcinoma. Transplantation. 2006 Jun 27;81(12):1633-9. doi: 10.1097/01.tp.0000226069.66819.7e. PMID 16794527
- [Background] Freeman RB, Mithoefer A, Ruthazer R, Nguyen K, Schore A, Harper A, Edwards E. Optimizing staging for hepatocellular carcinoma before liver transplantation: A retrospective analysis of the UNOS/OPTN database. Liver Transpl. 2006 Oct;12(10):1504-11. doi: 10.1002/lt.20847. PMID 16952174
- [Derived] Hoang MTQ, Koh YX, Sultana R, Allen JC, Moris D, Cheow PC, Chung AYF, Jeyaraj PR, Mack POP, Ooi LLPJ, Tan EK, Teo JY, Kam JH, Moe FNN, Chua JSS, Ng AWY, Goh JSQ, Goh BKP, Zani S, Chow PKH. Metroticket approach in a retrospective cohort study to predict overall survival after surgical resection for hepatocellular carcinoma. Int J Surg. 2024 Nov 1;110(11):7058-7066. doi: 10.1097/JS9.0000000000001868. PMID 39248314